CLINICAL TRIAL: NCT03809104
Title: Virtual Reality-based Rehabilitation in the Treatment and Prevention of Sarcopenia of Older Residents in Caring Facilities - a Pilot Study in Rural Southern Taiwan
Brief Title: VR-based Rehabilitation in the Treatment and Prevention of Sarcopenia of Older Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cishan Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Principal Investigator, Sheng-Hui Tuan, Attending Physician of Department of Rehabilitation, Cishan Hospital, Ministry of Health and Welfare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-034
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Sarcopenia
Keywords: virtual reality; sarcopenia; elderly
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: elder residents in caring facilities, including nursing home and daycare center 15 participants in nursing home and 15 participants in daycare center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- elderly with sarcopenia (Experimental): Virtual reality-based rehabilitation programs
  Interventions: Other: Virtual reality-based rehabilitation programs

INTERVENTIONS:
Other: Virtual reality-based rehabilitation programs — A virtual reality (VR)-based rehabilitation program that lasts for 12 weeks, twice per week, 30 minutes per time. The program was combined with progressive resistant training and functional movement of dominant upper (UE) limb. The device of the VR including one computer, one oculus headset, and one hand-hold sensor. The rehabilitation secession contains 4 different VR games in total, including (1) Leap Motion Blocks (2) Slum Ball VR Tournament (3) VR Super Sports 10th Edition- Basketball (4) VR Super Sports 10th Edition- Soccer.

SUMMARY:
Background:

Sarcopenia is the progressive loss of skeletal muscle mass and decline of muscle function associated with aging. The prevalence of sarcopenia among people older than 65 years old in Taiwan is over 20%. Sarcopenia is one of the most important causes of functional decline and loss of independence, even mortality in older adults. Literatures have found that resistant or aerobic exercise could improve muscle strength and function in older adults. However, due to shortage in healthcare provider, long-term rehabilitation program is difficult to provide in senior caring facilities of countryside in Taiwan.

Method:

The investigators conducted a study to screen sarcopenia among residents in senior caring facilities in Ci-Shan and Mei-Nong district, Kaohsiung, Taiwan. Older adults diagnosed as sarcopenia after screening received a virtual reality (VR)-based rehabilitation program that lasts for 12 weeks, twice per week, 30 minutes per time. The program was combined with progressive resistant training and functional movement of dominant upper (UE) limb. Criteria of sarcopenia including (1) handgrip strength of dominant hand (HGS), (2) walking speed, and (3) skeletal muscle mass of 4 extremities (SKM), were measured as primary outcomes. (1) Range of motions in dominant UE (ROM), (2) maximal voluntary isometric contraction of biceps/triceps brachial muscles of dominant side (MVC of biceps/triceps), and (3) box and block test (BBT), were measured as secondary outcomes before and after the programs.

Anticipated benefits:

VR-based rehabilitation program could enhance the motivation toward rehabilitation of older adults and reduce the health provider demand of senior caring facilities in countryside. It could also increase muscle mass, strength, and functional ability of dominant UE and reach the clinical effectiveness in treatment of sarcopenia.

DETAILED DESCRIPTION:
Sarcopenia is an involuntary loss of skeletal muscle mass and strength related with age. It is one of the most important causes of functional decline and loss of independence in older adults. In Taiwan, more than 20% of elders over the age of 65 are diagnosed with sarcopenia, and most of them are institutionalized. However, due to the lack of medical resources and medical professions, only a few elders with sarcopenia have received adequate rehabilitation. Recently, there are prevalence of research about integrating Virtual-Reality (VR) into various rehabilitations. Most of them have found that these VR-based rehabilitation can boost the motivation for participation, decrease the use of medical resources, and effectively contribute to the recovery of the patients. Inspired from these results, I think it might be interesting to integrate VR into the sarcopenia rehabilitation of elders.

This research has combined existed VR games with progressive resistance exercise of the upper limbs and exercises for the function movement system (F.M.S) of the upper limbs, establishing a VR-based rehabilitation program designed for sarcopenia elders. The rehabilitation programs spans for 8 weeks, and is conducted at least twice a week for each subject. The research question of this research is: "What is the impact of Virtual Reality-based rehabilitation on upper limb sarcopenia patient?".

The primary outcome of this research examines the change in muscle mass (measured by skeletal mass index, fat mass index and fat-free mass index), hand grip strength of the dominant hand and gait speed. The secondary outcome of this research examines the the change in range of motion of the upper limbs (shoulder flexion, shoulder external rotation, shoulder abduction, elbow flexion, elbow extension, elbow supination, elbow pronation, wrist flexion, wrist extension) and the functional ability of the upper limbs (measured by box and block test).

Hypothesis:

1. After two months of participating in the rehabilitation program, the primary outcomes (muscle mass, hand grip strength, and gait speed), show statistically significant increase.
2. After two months of participating in the rehabilitation program, the secondary outcomes (change of range of motion of the upper limbs and functional ability of upper limbs) show statistically significant increase.

Flow of the research:

1. Sarcopenia patients are first selected from the daycare and nursing home of Chi-Shan Hospital.
2. The first period of rehabilitation begins right after the selection and lasts for one month.
3. The first evaluation begins after the first period of rehabilitation
4. The second period of rehabilitation begins and lasts for one month.
5. The second evaluation begins after the second period of rehabilitation.

Apparatus in this study:

1. Leap Motion Controller
2. Oculus Rift headset (CV1)
3. Oculus Sensors (a pair)
4. (oculus) Touch Controllers
5. Omron KARADA Scan Body Composition & Scale (HBF-701)
6. JAMAR Hand Dynamometer
7. MicroFET3 Dynamometer and ROM Evaluator
8. Goniometer
9. Box and Block Test Apparatus

ELIGIBILITY:
Inclusion Criteria:

1. All the rehabilitation subjects are selected from the nursing home and day care center of Chi-Shan Hospital and over 60 years of age.
2. Participants meet the diagnostic criteria of sarcopenia based on the The Asian Working Group of Sarcopenia:

(1) Muscle mass lower than norm for two standard deviations and (2) Grip strength: men lower than 26 kg and women lower than 18 kg (measured by handgrip denominator used in physical examination) or an average gait speed lower than 0.8m/ sec.

3. Cognitive functions and physical strength are capable of completing the rehabilitation program which lasts for 30 minutes

Exclusion Criteria:

1. The ones who have uncontrollable high blood pressure, are recently infected, have major cardiovascular diseases and are prohibited to participate in sports exercise by the American College of Sports Medicine are excluded from the selection.
2. The ones who are bedridden are excluded from the selection.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cishan Hospital, Ministry of health and welfare, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ali S, Garcia JM. Sarcopenia, cachexia and aging: diagnosis, mechanisms and therapeutic options - a mini-review. Gerontology. 2014;60(4):294-305. doi: 10.1159/000356760. Epub 2014 Apr 8. PMID 24731978
- [Background] Frontera WR, Hughes VA, Fielding RA, Fiatarone MA, Evans WJ, Roubenoff R. Aging of skeletal muscle: a 12-yr longitudinal study. J Appl Physiol (1985). 2000 Apr;88(4):1321-6. doi: 10.1152/jappl.2000.88.4.1321. PMID 10749826
- [Background] Lexell J. Human aging, muscle mass, and fiber type composition. J Gerontol A Biol Sci Med Sci. 1995 Nov;50 Spec No:11-6. doi: 10.1093/gerona/50a.special_issue.11. PMID 7493202
- [Background] Janssen I, Heymsfield SB, Ross R. Low relative skeletal muscle mass (sarcopenia) in older persons is associated with functional impairment and physical disability. J Am Geriatr Soc. 2002 May;50(5):889-96. doi: 10.1046/j.1532-5415.2002.50216.x. PMID 12028177
- [Background] Janssen I, Shepard DS, Katzmarzyk PT, Roubenoff R. The healthcare costs of sarcopenia in the United States. J Am Geriatr Soc. 2004 Jan;52(1):80-5. doi: 10.1111/j.1532-5415.2004.52014.x. PMID 14687319
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Lo YC, Wahlqvist ML, Huang YC, Chuang SY, Wang CF, Lee MS. Medical costs of a low skeletal muscle mass are modulated by dietary diversity and physical activity in community-dwelling older Taiwanese: a longitudinal study. Int J Behav Nutr Phys Act. 2017 Mar 14;14(1):31. doi: 10.1186/s12966-017-0487-x. PMID 28288651
- [Background] Yarasheski KE, Pak-Loduca J, Hasten DL, Obert KA, Brown MB, Sinacore DR. Resistance exercise training increases mixed muscle protein synthesis rate in frail women and men >/=76 yr old. Am J Physiol. 1999 Jul;277(1):E118-25. doi: 10.1152/ajpendo.1999.277.1.E118. PMID 10409135
- [Background] Chen KM, Li CH, Chang YH, Huang HT, Cheng YY. An elastic band exercise program for older adults using wheelchairs in Taiwan nursing homes: a cluster randomized trial. Int J Nurs Stud. 2015 Jan;52(1):30-8. doi: 10.1016/j.ijnurstu.2014.06.005. Epub 2014 Jun 19. PMID 25037651
- [Background] Liu CJ, Latham NK. Progressive resistance strength training for improving physical function in older adults. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD002759. doi: 10.1002/14651858.CD002759.pub2. PMID 19588334
- [Background] Park DS, Lee DG, Lee K, Lee G. Effects of Virtual Reality Training using Xbox Kinect on Motor Function in Stroke Survivors: A Preliminary Study. J Stroke Cerebrovasc Dis. 2017 Oct;26(10):2313-2319. doi: 10.1016/j.jstrokecerebrovasdis.2017.05.019. Epub 2017 Jun 9. PMID 28606661
- [Background] Ilg W, Schatton C, Schicks J, Giese MA, Schols L, Synofzik M. Video game-based coordinative training improves ataxia in children with degenerative ataxia. Neurology. 2012 Nov 13;79(20):2056-60. doi: 10.1212/WNL.0b013e3182749e67. Epub 2012 Oct 31. PMID 23115212
- [Background] Garcia JA, Felix Navarro K, Schoene D, Smith ST, Pisan Y. Exergames for the elderly: towards an embedded Kinect-based clinical test of falls risk. Stud Health Technol Inform. 2012;178:51-7. PMID 22797019
- [Background] Bohannon RW. Test-retest reliability of the MicroFET 4 hand-grip dynamometer. Physiother Theory Pract. 2006 Sep;22(4):219-21. doi: 10.1080/09593980600822875. PMID 16920680
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Older adults aged more than 60 and lived in the nursing home or went to daycare center regularly in rural southern Taiwan were recruited for screening.All the residents with sufficient cognitive function and physical fitness to perform training that lasts for 30 minutes and meeting the criteria of sarcopenia by AWGS.
Pre-assignment Details: A total of 43 participants were recruited for VR-REH. Among them, 40 patients completed the study and 3 patients withdrew during the study period (2 dropped out during the visit at 4 weeks due to hospitalization and 1 withdrew at 8 weeks due to case-closed from daycare center).
Period: Overall Study
Arm/Group | Elderly With Sarcopenia
Started | 43
Completed | 40
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Elderly With Sarcopenia
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.57 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 40
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — A total of 43 participants were recruited initially. Among them, 40 patients completed the study and 3 patients withdrew during the study period (2 dropped out before the 4th week due to hospitalization and 1 withdrew before the 4th week due to case-closed from daycare center). Therefore, the data we measured and analyzed were all from the 40 patients who completed the study.
  participants
    Taiwan | 40
Height [Mean (Standard Deviation); unit: cm] | 156.97 (8.76)
Weight [Mean (Standard Deviation); unit: kg] | 58.74 (10.89)

OUTCOME MEASURES:

1. Primary Outcome: Change of Hand-grip Strength of the Dominant Hand Between the Third Month and the Baseline
Description: The measurements of the HGS were determined by means of the JAMAR-Dynamometer. The forearm was held in neutral position and the wrist at a 0 to 30° extension. The instrument was held freely: neither the hand nor the forearm was allowed to rest on a surface. Three measurements were done and recorded as the average of the three measurements and the participants rested for 1 minute in between measurements.
  The change was calculated by the data of the third month minus the baseline data.
Time Frame: 3 months after the intervention of the virtual reality-based rehabilitation programs
Measure: Median (Standard Deviation); unit: kg
Arm/Group | Elderly With Sarcopenia
Number analyzed (Participants) | 40
kg | 5.02 (1.25)

2. Primary Outcome: Change of Walking Speed Between the Third Month and the Baseline
Description: Timing starts after the patient starts walking and stops at the point when a patient reaches a distance of 6 meters. The gait speed in measured twice and the final measurement is the average of the two scores. The patient is allowed to rest for 10 minutes in between measurement.
  The change was calculated by the data of the third month minus the baseline data.
Time Frame: 3 months after the intervention of the virtual reality-based rehabilitation programs
Measure: Mean (Standard Deviation); unit: meter/second
Arm/Group | Elderly With Sarcopenia
Number analyzed (Participants) | 40
meter/second | 0.2 (0.06)

3. Primary Outcome: Change of Appendicular Skeletal Muscle Mass Between the Third Month and the Baseline
Description: Appendicular skeletal muscle mass (ASM) is deﬁned by the sum of the lean soft tissue mass of four limbs. Appendicular skeletal muscle mass index (ASMI) is defined as ASM (kg) divided by squared height (m).The body composition was measured via bio-electrical impedance analysis by Omron KARADA Scan Body Composition & Scale (HBF-701). A participant was considered to have low muscle mass if his or her ASMI was below -2 standard deviations of the reference defined in previous studies from Taiwan (6.76 kg/m2 for men and 5.28 kg/m2 for women). Participants with ASMI in the lowest 20% of the sex-specific distribution were considered to have low muscle mass, too. Increased of ASMI after virtual reality-based rehabilitation programs is considered to be better.
  The change was calculated by the data of the third month minus the baseline data.
Time Frame: 3 months after the intervention of the virtual reality-based rehabilitation programs
Measure: Mean (Standard Deviation); unit: kg/meter square
Arm/Group | Elderly With Sarcopenia
Number analyzed (Participants) | 40
kg/meter square | 0.21 (0.06)

4. Secondary Outcome: Range of Motions in Dominant Upper Extremity
Description: Use goniometry for range of motion measurement. The joints measured include shoulder, elbow, and wrist of the dominant side.
Time Frame: baseline;1, 2, and 3 months after the intervention of the virtual reality-based rehabilitation programs
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Elderly With Sarcopenia
Number analyzed (Participants) | 40
degree
  shoulder flexion (baseline) | 130.36 (14.32)
  shoulder flexion (the first month) | 139.07 (11.01)
  shoulder flexion (the second month) | 143.07 (8.43)
  shoulder flexion (the third month) | 149.79 (8.70)
  shoulder external rotation (baseline) | 71.68 (10.64)
  shoulder external rotation (the first month) | 75.50 (5.95)
  shoulder external rotation (the second month) | 77.36 (4.68)
  shoulder external rotation (the third month) | 79.50 (3.70)
  shoulder abduction (baseline) | 128.79 (25.61)
  shoulder abduction (the first month) | 130.71 (15.70)
  shoulder abduction (the second month) | 138.21 (9.94)
  shoulder abduction (the third month) | 141.93 (9.82)
  elbow flexion (baseline) | 120.29 (10.89)
  elbow flexion (the first month) | 117.29 (7.57)
  elbow flexion (the secondt month) | 118.79 (8.54)
  elbow flexion (the third month) | 119.93 (6.88)
  elbow extension (baseline) | 3.71 (2.77)
  elbow extension (the first month) | 3.43 (1.55)
  elbow extension (the second month) | 3.79 (1.12)
  elbow extension (the third month) | 4.64 (0.63)
  elbow supination (baseline) | 56.07 (15.27)
  elbow supination (the first month) | 56.64 (9.95)
  elbow supination (the second month) | 59.14 (9.24)
  elbow supination (the third month | 66.86 (9.45)
  elbow pronation (baseline) | 59.43 (18.33)
  elbow pronation (the first month) | 60.43 (13.23)
  elbow pronation (the second month) | 63.21 (13.10)
  elbow pronation (the third month) | 69.21 (9.37)
  wrist flexion (baseline) | 51.86 (9.80)
  wrist flexion (the first month) | 56.36 (8.82)
  wrist flexion (the second month) | 62.07 (5.90)
  wrist flexion (the third month) | 66.71 (4.68)
  wrist extension (baseline) | 52.50 (10.90)
  wrist extension (the first month) | 58.64 (12.60)
  wrist extension (the second month) | 65.93 (9.04)
  wrist extension (the third month) | 69.86 (7.49)

5. Secondary Outcome: Strength of Biceps Brachii and Triceps Brachii of the Dominant Upper Extremity
Description: This research uses MicroFET3 to measure the the maximal voluntary isometric contraction of the biceps and triceps. Measurements are taken 2 times and the results are averaged. MicroFET3 is a electronic hand-held dynamometer that can measure muscle strength. The range of muscle testing of the device ranges from 0-150 lbs force.(Digital Dynamometer and Inclinometer | MicroFET®3) .
Time Frame: baseline;1, 2, and 3 months after the intervention of the virtual reality-based rehabilitation programs
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Elderly With Sarcopenia
Number analyzed (Participants) | 40
kg
  Strength of biceps brachii muscle (baseline) | 5.03 (1.31)
  Strength of biceps brachii muscle (the 1st month) | 5.48 (1.28)
  Strength of biceps brachii muscle (the 2nd month) | 5.80 (1.22)
  Strength of biceps brachii muscle (the 3rd month) | 6.44 (1.21)
  Strength of triceps brachii muscle (baseline) | 5.06 (1.20)
  Strength of triceps brachii muscle (the 1st month) | 5.55 (1.35)
  Strength of triceps brachii muscle (the 2nd month) | 5.75 (1.12)
  Strength of triceps brachii muscle (the 3rd month) | 6.15 (1.27)

6. Secondary Outcome: Box and Block Test
Description: The Box and Block Test (BBT) can measure the unilateral gross manual dexterity. The set up of the BBT test includes a wooden box with 150 wooden blocks inside. The wooden box is divided into two compartments. One filled with blocks, and the other is empty.During this test, the patient is seated upright in a chair and needs to transfer the wooden blocks, one by one, from one compartment to the other. The patient is scored based on the number of blocks he or she can transferred from one compartment to the other in 60 seconds.
Time Frame: baseline;1, 2, and 3 months after the intervention of the virtual reality-based rehabilitation programs
Measure: Mean (Standard Deviation); unit: boxes
Arm/Group | Elderly With Sarcopenia
Number analyzed (Participants) | 40
boxes
  number (baseline) | 26.86 (12.63)
  number (the first month) | 34.14 (13.12)
  number (the second month) | 36.04 (9.31)
  number (the third month) | 37.57 (12.91)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Elderly With Sarcopenia
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 8/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elderly With Sarcopenia (N=40)
light-headedness (Ear and labyrinth disorders) | 5 (5) — The symptom presented at the last 20 minutes of each session of the program and it subsided after stopping the virtual reality device.
sore eyes (Eye disorders) | 3 (3) — the symptom developed after the 30-minute VR-based program and it resolved after resting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-12-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT03809104/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT03809104/SAP_001.pdf